CLINICAL TRIAL: NCT00480727
Title: Determining Optimal Halo Pin Management Practises to Decrease Pin Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 135/07; A10704
Record Dates: First submitted 2007-05-29; First posted 2007-05-31 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2010-05

CONDITIONS: Unstable Cervical Injury
Keywords: Halo Thoracic Orthosis; Re-tension; Pin loosening

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): No fortnightly re-tensioning. Placebo treatment utilises the re-tensioning procedure, pt experiences clicking sensation, however, the pin is not tightened.
  Interventions: Procedure: Placebo Re-tensioning
- Treatment (Re-tensioning) Group (Experimental): Pins are re-tensioned fortnightly back to initial fitting tension of 8lb/inch.
  Interventions: Procedure: Halo pin re-tensioning

INTERVENTIONS:
Procedure: Halo pin re-tensioning — Re-tensiong every 2 weeks with torque driver. Pins are re-tensioned to 8lb/inch
  Arms: Treatment (Re-tensioning) Group
Procedure: Placebo Re-tensioning — Pts undergo re-tensioning procedure with torque driver set at zero to elicit the same clicking sensation with no tightening of the pin.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effects of regular pin re-tensioning on pain, pin loosening and pin replacement.

DETAILED DESCRIPTION:
Halo Thoracic Orthoses (Halos) are used to immobilise unstable cervical fractures. The halo grips the skull via 4 pins. Pin loosening is a major complication of halo wear. Pin loosening is painful and can result in loss of control of the fractures. Treatment is required urgently and involves re-siting the pin.

Comparisons: This study will compare two pin management practises with the aim to determine which is optimal to reduce the incidence of complications including pin loosening. Patients will be randomly allocated into 2 groups. The control group will receive treatment in accordance with current practise at The Alfred, the pins will not be re-tensioned throughout the treatment period. The alternative treatment group will have their pins re-tensioned fortnightly.

ELIGIBILITY:
Inclusion Criteria:

* Must be fitted with a Halo Thoracic Orthosis at The Alfred Hospital

Exclusion Criteria:

* Patients who can not have their halo pins tensioned to at least 8lb/inch pressure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Pin Complications | Treatment duration (approx 12 weeks)
  Pins classified at each follow-up as OK, At Risk, Loose, Moderate or Severe Infection

SECONDARY OUTCOMES:
Anxiety Text | Fortnightly
Pain | Fortnightly
  Pain measured on a numerical rating scale 0-10 at each review both before and after treatment is provided
Pin Tension Measurements | Fornightly
  Pin tensioned measured fortnightly using torque reading device

CONTACTS AND LOCATIONS:
Overall Officials: Karly N Wheeler, Bach Prosthetics & Orthotics, Principal Investigator — The Alfred Hospital, Bayside Health
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Background] Kuester WM, Stamper RE, Ordway NR. Analysis of pin force distributions of halo orthoses. Biomed Sci Instrum. 2002;38:221-6. PMID 12085606
- [Background] Garfin SR, Botte MJ, Waters RL, Nickel VL. Complications in the use of the halo fixation device. J Bone Joint Surg Am. 1986 Mar;68(3):320-5. PMID 3949826
- [Background] Vertullo CJ, Duke PF, Askin GN. Pin-site complications of the halo thoracic brace with routine pin re-tightening. Spine (Phila Pa 1976). 1997 Nov 1;22(21):2514-6. doi: 10.1097/00007632-199711010-00010. PMID 9383858